CLINICAL TRIAL: NCT04802967
Title: A Phase I, Double-Blind, PK, Safety, Tolerability Study of KSL + KLS-GABA vs KLS Alone in Healthy Males (Part A) Followed by a Study to Investigate the PD of KLS and KLS + GABA in Healthy Males (Part B)
Brief Title: A Study on Ketoprofen Lysine Salt (KLS) + Gabapentin (GABA) vs KLS to Investigate Their Pharmacodynamic in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KLG0120; 2020-004212-10 (EudraCT Number)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: No Condition
Keywords: Male healthy volunteers
MeSH Terms: interventions — Gabapentin; gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: In the Part B of the study the Intradermal (ID) Capsaicin Model is used.
Who Masked: Participant, Investigator
Masking Description: This study will be double-blinded (Investigator- and subject-blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KLS-GABA (part A and B) (Experimental): KLS-GABA 80 mg-34 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomisation schedule. Capsules are administered with 240 mL of water.
  KLS-GABA (40 mg-17mg, 80 mg-34 mg, or 160 mg-68 mg) in Part B are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water.
  To maintain he blind, subjects assigned to receive 160 mg-68 mg KLS-GABA are administered two co-crystal KLS-GABA 114 mg (80 mg-34 mg) capsules, and subject assigned to receive 40 mg-17 mg KLS-GABA or 80 mg-34 mg KLS-GABA also receive a placebo capsule (dummy placebo).
  Interventions: Drug: Ketoprofen Lysine Salt combined with Gabapentin
- KLS (part A and B) (Active Comparator): KLS 80 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomisation schedule. Capsules will be administered with 240 mL of water.
  In the part B KLS (40 mg, 80 mg or 160 mg) are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water. To maintain the blind, subjects assigned to receive 160 mg KLS alone are administered two KLS 80 mg capsules and subjects assigned to receive either 40 mg KLS alone or 80 mg KLS alone also receive a placebo capsule (dummy placebo).
  Interventions: Drug: Ketoprofen Lysine Salt
- Gabapentin (part B) (Active Comparator): Gabapentin 300 mg are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water.To maintain the blind, subjects assigned to receive 300 mg gabapentin also receive a placebo capsule (dummy placebo).
  Interventions: Drug: Gabapentin
- Placebo (part B) (Placebo Comparator): To maintain the blind subjects assigned to receive placebo receive 2 placebo capsules. Capsules will be administered with 240 mL of water.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketoprofen Lysine Salt combined with Gabapentin — KLS-GABA (80 mg-34 mg) in Part A and KLS-GABA (40 mg-17 mg or 80 mg-34 mg or 160 mg-68 mg) in Part B
  Other Names: KLS-GABA
  Arms: KLS-GABA (part A and B)
Drug: Ketoprofen Lysine Salt — KLS (80 mg) alone in each treatment period in Part A and KLS alone (40 mg, 80 mg, or 160 mg) in Part B
  Other Names: KLS
  Arms: KLS (part A and B)
Drug: Gabapentin — 300 mg
  Other Names: GABA
  Arms: Gabapentin (part B)
Other: Placebo — 2 capsules to maintain the blind
  Arms: Placebo (part B)

SUMMARY:
Part A The primary objective of this study is to determine the single dose pharmacokinetics (PK) of ketoprofen lysine salt combined with gabapentin (KLS-GABA [80 mg-34 mg]) compared to KLS alone (80 mg) in healthy male subjects.

The secondary objective of this study is:

• To determine the safety and tolerability of a single oral dose of KLS-GABA (80 mg-34 mg) compared to KLS alone (80 mg) in healthy male subjects.

Part B The primary objective of this study is to determine the pharmacodynamic (PD) effects of KLS-GABA in the Intradermal (ID) capsaicin model in healthy male subjects.

The secondary objectives of this study are:

* To further investigate the safety, tolerability, and PK of single oral doses of KLS-GABA and KLS alone.
* To investigate the possible relationship between plasma levels of drug and efficacy in pain reduction.

DETAILED DESCRIPTION:
This is a Phase I, Double-Blind, Pharmacokinetic, Safety and Tolerability Study of Ketoprofen Lysine Salt Combined with Gabapentin (KLS-GABA) Compared to Ketoprofen Lysine Salt (KLS) Alone in Healthy Male Subjects (Part A) Followed by a Randomised, Double-Blind, Placebo-Controlled Study to Investigate the Pharmacodynamic Effects of KLS, and KLS in Combination with Gabapentin (GABA), in Healthy Male Subjects Using the Intradermal (ID) Capsaicin Model (Part B).

Part A is a randomized, double-blind, crossover group study to investigate the safety, tolerability, and PK profile of a single oral dose of KLS-GABA compared to KLS alone in healthy male subjects. It is planned to enroll 12 subjects. All subjects take part in 2 treatment periods, in which they are randomized to receive either a single dose of KLS-GABA (80 mg-34 mg) or a single dose of KLS (80 mg) alone in each treatment period.

Subjects' participation in Part A lasts approximately 7 weeks and will consist of the following:

* A screening visit (up to 28 days prior to Day 1 of Treatment Period 1),
* Admission to the clinical research unit (CRU) on Day -1 prior to Treatment Period 1,
* Treatment Period 1 (Day 1 to Day 3),
* A washout period of a minimum of 7 days,
* Admission to the CRU on Day -1 prior to Treatment Period 2,
* Treatment Period 2 (Day 1 to Day 3),
* A follow-up visit (5 to 7 days post-final dose following Treatment Period 2). Safety will is assessed through Adverse Events (AE) reporting, 12-lead ECGs, vital signs, physical examinations, and clinical laboratory examinations. Pharmacokinetics are assessed by blood sampling.

Part A treatment lasts 2 days (Day 1 in Treatment Period 1; Day 1 in Treatment Period 2)

Part B is a randomized, double-blind, placebo-controlled parallel-group study to investigate the PD effects, PK/PD correlation, safety, and tolerability of three single oral dose levels of KLS-GABA compared to KLS alone, 300 mg gabapentin and placebo in the ID capsaicin model in healthy male subjects.

It is planned to enroll 128 subjects, randomized evenly to 8 possible treatments; subjects receive either KLS alone, KLS-GABA, 300 mg gabapentin or placebo. The planned treatments are:

* KLS alone (40 mg, 80 mg, or 160 mg)
* KLS-GABA (40 mg-17 mg, 80 mg-34 mg or 160 mg-68 mg)
* Gabapentin (300 mg)
* Placebo

Subjects' participation in Part B lasts approximately 6 weeks and consists of the following:

* A screening visit (up to 28 days prior to dosing)
* An additional screening visit (at least 7 days prior to dosing) to determine the subject's response to capsaicin and to familiarise them in the pain measurements,
* Admission to the CRU on Day -1, for collection of pain measurements and completion of the ID capsaicin model
* A treatment period (morning of Day 1 until 12 hours postdose)
* Discharge from the CRU 12 hours postdose
* A follow-up visit (5 to 7 days postdose). Safety is assessed through AE reporting, 12-lead ECGs, vital signs, physical examinations, and clinical laboratory examinations. Pharmacokinetics are assessed by blood sampling. Pharmacodynamics are assessed using the ID capsaicin model and pain measurements. Part B treatment lasts 1 day (Day 1).

ELIGIBILITY:
Inclusion Criteria:

Part A

Subjects meeting the following criteria will be included in the study:

1. Subject is male, of any ethnic origin.
2. Subject is aged between 18 to 55 years, inclusive.
3. Subject has a body mass index (BMI) of 18 to 32 kg/m2, inclusive.
4. Subject is ≥50 kg.
5. Negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test at Screening and Day -1 in each treatment period.
6. Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examinations, concomitant medication, vital signs, 12-lead ECG, and clinical laboratory evaluations.
7. Subjects must use a condom during the trial and for 3 months after their final dose of trial medication, if their partner is a woman of childbearing potential. In addition, their female partner of childbearing potential must use an additional method of highly effective contraception (see Section 6.4.1) from dosing until 3 months following dosing.
8. Subject is either a non-smoker or does not smoke more than 5 cigarettes per day (or equivalent e-cigarette use).
9. Provision of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Part B

Subjects meeting the following criteria will be included in the study:

1. Subject is male, with a skin type compatible with capsaicin measurements.
2. Subject is aged between 18 to 55 years, inclusive.
3. Subject has a BMI of 18 to 32 kg/m2, inclusive.
4. Subject is ≥50 kg.
5. Negative SARS-CoV-2 test at Screening and Day -1.
6. Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examination, concomitant medication, vital signs, 12-lead ECG, and clinical laboratory evaluations.
7. Subject must be in good general health with a skin type compatible with the measures, and without significant skin allergies, pigmentary disorders, or any active dermatological conditions that might interfere with the conduct of the study.
8. Subjects must use a condom during the trial and for 3 months after their final dose of trial medication, if their partner is a woman of childbearing potential. In addition, their female partner of childbearing potential must use an additional method of highly effective contraception (see Section 6.4.1) from dosing until 3 months following dosing.
9. Subjects must be able to tolerate the capsaicin injection at screening.
10. Demonstration of positive hyperalgesia as defined by an area of hyperalgesia ≥15 cm2 15 minutes after ID administration of 100 μg capsaicin at the additional screening visit at least 7 days prior to first dosing.
11. Subject is a either non-smoker or does not smoke more than 5 cigarettes per day (or equivalent e-cigarette use).
12. Provision of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

Part A

Subjects with any of the following will be excluded from study participation:

1. Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations obtained during screening as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine/diabetic, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder).
2. Clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), 12-lead ECG and vital signs, or physical findings at screening. In case of uncertain or questionable results, tests performed during screening may be repeated once to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
3. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism and excretion (ADME) of the study drugs.
4. Any other concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study as outlined in this Protocol, safety of the subject as per the SmPC of KLS and gabapentin (Neurontin 300 mg hard capsules) or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
5. Subject has a history of neurological disorders which may impact the perception of pain or impairs the subject's ability to fully participate in the study.
6. Subject has a significant skin allergy, pigmentary disorder, or any active dermatological condition.
7. AST, ALT, gamma-glutamyl transferase (GGT) or total bilirubin levels above the ULN at screening. These laboratory evaluations may be repeated once at the discretion of the Investigator. If the repeat test is within the reference range, the subject may be included only if the Investigator considers that the previous finding will not introduce additional risk factors and will not interfere with interpretation of safety data.
8. Positive test for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibody (anti- HCV) or human immunodeficiency virus I and II antibodies (anti-HIV I/II) at screening.
9. Positive urine test for drugs of abuse or alcohol breath test at screening or Day -1 of each treatment period.
10. History of drug and/or alcohol abuse/dependence, or intake of >28 units of alcohol weekly, and the inability to refrain from alcohol use from 48 hours before screening and each scheduled visit until discharge from the CRU. One unit is equivalent to a 285 mL glass of full strength beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine.
11. Habitual and heavy consumption of caffeinated beverages (>8 cups of coffee or equivalent per day) at screening; and/or unable to refrain from use of (methyl) xanthine (e.g., coffee, tea, cola, chocolate) from 48 hours prior to dosing until discharge from the CRU.
12. The subject has participated in a clinical study and has received a medication or a new chemical entity within 3 months or 5 half-lives (whichever is longer) prior to dosing of current study medication.
13. Use of any prescription or non-prescription medications, including herbal and nutritional supplements (including St. John's wort), or OTC medications (e.g., ibuprofen, aspirin) within 14 days of dosing and throughout the study. By exception, the subject may take acetaminophen (less or equal 2 g/day) for up to 48 hours prior to dosing. The Investigator and study team may review medication on a case-by-case basis to determine if its use would compromise subject safety or interfere with study procedures or data interpretation.
14. History of severe adverse reactions or allergies, or history of an anaphylactic reaction to prescription medications, non-prescription medication, food, NSAIDs or gabapentin (non-active hay-fever is acceptable).
15. Consumption of any food or drinks containing cranberry, pomegranate, starfruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges (including marmalade and juices made from these fruits) within 14 days before admission to the CRU until the end of the study.
16. Strenuous exercise within 48 hours prior to each blood collection for clinical laboratory tests.
17. Donation of blood or plasma of >500 mL within 3 months prior to first dosing, or subject intends to donate blood during the study.
18. Male subject who will not abstain from sperm donation between dosing and 3 months after final dosing.
19. Any degree of previous or known hypersensitivity to the active substance or the excipients of the IMP.

Part B

Subjects with any of the following will be excluded from study participation:

1. Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations obtained during screening as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine/diabetic, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder).
2. Clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), 12-lead ECG and vital signs, or physical findings at screening. In case of uncertain or questionable results, tests performed during screening may be repeated once to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
3. Has a skin trauma, any active skin disorder, significant scarring, significant skin allergy, pigmentary disorder, active dermatological condition, skin disease or tattoos on either forearm, or a significant history of trauma or skin disease in either arm.
4. Subject has a known intolerance to capsaicin, hot peppers, or any excipient in the IMP.
5. Subject has active chronic pain condition(s) or a history of chronic pain conditions.
6. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the ADME of the study drug.
7. Any other concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study as outlined in this Protocol, safety of the subject as per the SmPCs of KLS and gabapentin (Neurontin 300 mg hard capsules) or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
8. Subject has a history of neurological disorders which may impact the perception of pain or impairs the subject's ability to fully participate in the study.
9. AST, ALT, GGT or total bilirubin levels above the ULN at screening. These laboratory evaluations may be repeated once at the discretion of the Investigator. If the repeat test is within the reference range, the subject may be included only if the Investigator considers that the previous finding will not introduce additional risk factors and will not interfere with interpretation of safety data.
10. Positive test for HBsAg, anti-HCV or anti-HIV I/II at screening.
11. Positive urine test for drugs of abuse or alcohol breath test at screening.
12. History of drug and/or alcohol abuse/dependence, or intake of >28 units of alcohol weekly, and the inability to refrain from alcohol use from 48 hours before Screening and each scheduled visit until discharge from the CRU. One unit is equivalent to a 285 mL glass of full strength beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine.
13. Habitual and heavy consumption of caffeinated beverages (>8 cups of coffee or equivalent per day) at screening; and/or unable to refrain from use of (methyl) xanthine (e.g., coffee, tea, cola, chocolate) from 48 hours prior to dosing until discharge from the CRU.
14. The subject has participated in a clinical study and has received a medication or a new chemical entity within 3 months or 5 half-lives (whichever is longer) prior to dosing of current study medication.
15. Use of any prescription or non-prescription medications, including herbal and nutritional supplements (including St. John's wort), or OTC medications (e.g., ibuprofen, aspirin) within 14 days of dosing and throughout the study. By exception, the subject may take acetaminophen (less or equal 2 g/day) for up to 48 hours prior to dosing. The Investigator and study team may review medication on a case-by-case basis to determine if its use would compromise subject safety or interfere with study procedures or data interpretation.
16. History of severe adverse reactions or allergies, or history of an anaphylactic reaction to prescription medication, non-prescription medication, food, NSAIDs, gabapentin, (non-active hay-fever is acceptable), the planned local anaesthesia/analgesic regimens, ethylenediaminetetraacetic acid, Kolliphor HS 15, butylated hydroxytoluene, or capsaicin.
17. Known hypersensitivity or allergy to any component of the placebo capsules.
18. Consumption of any food or drinks containing cranberry, pomegranate, starfruit, grapefruit, pomelos, exotic citrus fruits, or Seville oranges (including marmalade and juices made from these fruits) within 14 days before admission to the CRU until the end of the study.
19. Strenuous exercise within 48 hours prior to each blood collection for clinical laboratory tests.
20. Subject has participated in a clinical study involving administration of capsaicin within 12 months of the screening visit.
21. Donation of blood or plasma of >500 mL within 3 months prior to dosing, or subject intends to donate blood during the study.
22. Male subject who will not abstain from sperm donation between dosing and 3 months after dosing.
23. Any degree of previous or known hypersensitivity to the active substance or the excipients of the IMP.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subject is male, of any ethnic origin. Subject is aged between 18 to 55 years, inclusive. Subject has a body mass index (BMI) of 18 to 32 kg/m2, inclusive and ≥50 kg.
Enrollment: 141 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pui Man Leung, BMChB, MRCP, Principal Investigator — MAC Clinical Research Early Phase Unit
Locations (1):
- MAC Clinical Research Early Phase Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: "Enrolled" is any subject who signed an ICF. "Randomized" are patients randomly assigned evenly between treatment sequences; "Dosed" is any subject who actually received at least one dose of IMP during the relevant Part.
  In part A: n= 6 for all these definitions. In Part B: the enrolled and randomized were n=129; the dosed population is n=128 because 1 pt was randomized to the KLS 40 mg-GABA 17 mg but withdrawn prior to dosing due to a code break issue.
Pre-assignment Details: Separate randomization schemes were produced for each Part A (cross-over) of the study and Part B of the study. A simple randomization scheme was used for Part A, while a blocked randomization scheme was used for Part B.
  Please note: Given the differences between Part A and Part B (design, objectives, endpoints, etc.) study results of the two parts cannot be merged.
Groups:
- "KLS 80 mg Alone, *Then* KLS 80 Mg and GABA 34 mg" (PART A); "KLS 80 Mg and GABA 34 mg *Then* KLS 80 mg Alone" (PART A): KLS-GABA 80 mg-34 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules are administered with 240 mL of water.
  To maintain the blind, subjects assigned to receive 80 mg-34 mg KLS-GABA also receive a placebo capsule (dummy placebo).
  KLS 80 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules will be administered with 240 mL of water.
  Ketoprofen Lysine Salt combined with Gabapentin: KLS-GABA (80 mg-34 mg) in Part A Ketoprofen Lysine Salt: KLS (80 mg) alone in each treatment period in Part A
- KLS 40 mg; KLS 80 mg; KLS 160 mg: In the part B KLS (40 mg, 80 mg or 160 mg) are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water. To maintain the blind, subjects assigned to receive 160 mg KLS alone are administered two KLS 80 mg capsules and subjects assigned to receive either 40 mg KLS alone or 80 mg KLS alone also receive a placebo capsule (dummy placebo).
- KLS 40 Mg-GABA 17 mg; KLS 80 mg- GABA 34 mg; KLS 160 Mg-GABA 68 mg: KLS-GABA (40 mg-17mg, 80 mg-34 mg, or 160 mg-68 mg) in Part B are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water.
  Subject assigned to receive 40 mg-17 mg KLS-GABA or 80 mg-34 mg KLS-GABA also receive a placebo capsule (dummy placebo).
- Gabapentin 300 mg: Gabapentin 300 mg are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water.To maintain the blind, subjects assigned to receive 300 mg gabapentin also receive a placebo capsule (dummy placebo).
- Placebo: To maintain the blind subjects assigned to receive a placebo receive 2 placebo capsules. Capsules will be administered with 240 mL of water.
  Placebo: 2 capsules to maintain the blind
Period: Part A
Arm/Group | "KLS 80 mg Alone, *Then* KLS 80 Mg and GABA 34 mg" (PART A) | "KLS 80 Mg and GABA 34 mg *Then* KLS 80 mg Alone" (PART A) | KLS 40 mg | KLS 80 mg | KLS 160 mg | KLS 40 Mg-GABA 17 mg | KLS 80 mg- GABA 34 mg | KLS 160 Mg-GABA 68 mg | Gabapentin 300 mg | Placebo
Started | 6 (This group participates only in part A) | 6 (This group participates only in part A) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B)
Enrolled, Randomized and Dosed (Enrolled is any subject who signed an informed consent form.) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 (This group participates only in part A) | 6 (This group participates only in part A) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B) | 0 (This group participates only in part B)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | "KLS 80 mg Alone, *Then* KLS 80 Mg and GABA 34 mg" (PART A) | "KLS 80 Mg and GABA 34 mg *Then* KLS 80 mg Alone" (PART A) | KLS 40 mg | KLS 80 mg | KLS 160 mg | KLS 40 Mg-GABA 17 mg | KLS 80 mg- GABA 34 mg | KLS 160 Mg-GABA 68 mg | Gabapentin 300 mg | Placebo
Started | 0 (This group participates only in part A) | 0 (This group participates only in part A) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 17 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B)
Enrolled, Randomized and Dosed (Overall, in part B, 129 subjects were enrolled and 128 were dosed during Part B of the study, because 1 pt withdrawn prior to dosing due to a code break issue. All the 128 subjects dosed were randomised evenly across treatment groups and completed Part B of the study.) | 0 | 0 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
Completed | 0 (This group participates only in part A) | 0 (This group participates only in part A) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B) | 16 (This group participates only in part B)
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Analysis Set consisted of all subjects randomized. A subject's randomized treatment sequence was used for analysis regardless of the actual treatment received. Please note: Given the differences between Part A and Part B (design, objectives, endpoints, etc.) as per study design, the first two columns, pertaining to PART A, are given per sequence and not per arm.
  .
Groups:
- KLS 40 mg (Part B); KLS 80 mg (Part B); KLS 160 mg (Part B): In the part B KLS (40 mg, 80 mg or 160 mg) are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water. To maintain the blind, subjects assigned to receive 160 mg KLS alone are administered two KLS 80 mg capsules and subjects assigned to receive either 40 mg KLS alone or 80 mg KLS alone also receive a placebo capsule (dummy placebo).
- KLS 40 Mg-GABA 17 mg (Part B); KLS 80 mg- GABA 34 mg (Part B); KLS 160 Mg-GABA 68 mg (Part B): KLS-GABA (40 mg-17mg, 80 mg-34 mg, or 160 mg-68 mg) in Part B are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water.
  Subject assigned to receive 40 mg-17 mg KLS-GABA or 80 mg-34 mg KLS-GABA also receive a placebo capsule (dummy placebo).
- Gabapentin 300 mg (Part B): Gabapentin 300 mg are administered as capsules once in the morning of Day 1 in the fasted state. Capsules are administered with 240 mL of water.To maintain the blind, subjects assigned to receive 300 mg gabapentin also receive a placebo capsule (dummy placebo).
  Gabapentin: 300 mg
- Placebo (Part B): To maintain the blind subjects assigned to receive a placebo receive 2 placebo capsules. Capsules will be administered with 240 mL of water.
  Placebo: 2 capsules to maintain the blind
- Total: Total of all reporting groups
Arm/Group | "KLS 80 mg Alone, *Then* KLS 80 Mg and GABA 34 mg" (PART A) | "KLS 80 Mg and GABA 34 mg *Then* KLS 80 mg Alone" (PART A) | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B) | Total
Number analyzed (Participants) | 6 | 6 | 16 | 16 | 16 | 17 | 16 | 16 | 16 | 16 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 16 | 16 | 16 | 17 | 16 | 16 | 16 | 16 | 141
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (4.93) | 29.5 (10.43) | 29.3 (8.23) | 30.8 (12.86) | 28.1 (10.39) | 29.2 (8.92) | 31.1 (9.68) | 27.1 (9.57) | 27.1 (10.51) | 28.9 (10.01) | 29.0 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 16 | 16 | 16 | 17 | 16 | 16 | 16 | 16 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 4 | 5 | 15 | 16 | 15 | 17 | 16 | 14 | 15 | 16 | 133
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 16 | 16 | 16 | 17 | 16 | 16 | 16 | 16 | 141

OUTCOME MEASURES:

1. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): Area Under the Concentration-time Curve (AUC) From Zero to the Last Quantifiable Concentrations (AUC0-t),
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  Outcome measure at 0h,16h,24h,36h, and 48h postdose below limit of quantification (0.04 μg/mL).
  The area under the concentration versus time curve from time zero to the last quantifiable concentration (C-last), calculated by the linear up-log down trapezoidal method; i.e. when concentrations are increasing (as in the absorption phase), the linear trapezoidal method is used, when concentrations are decreasing (as in the elimination phase), the logarithmic trapezoidal method is used.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Groups:
- KLS 80 mg (Part A): KLS 80 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules will be administered with 240 mL of water.
- KLS 80 Mg-GABA 34 mg (Part A): KLS-GABA 80 mg-34 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules are administered with 240 mL of water.
  To maintain the blind, subjects assigned to receive 80 mg-34 mg KLS-GABA also receive a placebo capsule (dummy placebo).
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
μg*h/mL | 10.5 (2.70) | 11.1 (2.94)

2. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A):AUC From Zero to 12 Hours Postdose (AUC0-12h)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  The area under the concentration versus time curve from time zero to 12 h post-dose, calculated by the linear up-log down trapezoidal method.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
μg*h/mL | 10.3 (2.25) | 11.0 (2.89)

3. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): AUC From Zero to 24 Hours Postdose (AUC0-24h)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  The area under the concentration versus time curve from time zero to 24 h post-dose, calculated by the linear up-log down trapezoidal method.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
μg*h/mL | 10.5 (2.42) | 11.2 (3.02)

4. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A):AUC From Zero to 36 Hours Postdose (AUC0-36h)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.The area under the concentration versus time curve from time zero to 36 h post-dose, calculated by the linear up-log down trapezoidal method.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
μg*h/mL | 10.5 (2.56) | 11.2 (3.00)

5. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): AUC From Zero to 48 Hours Postdose (AUC0-48h)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.The area under the concentration versus time curve from time zero to 48 h post-dose, calculated by the linear up-log down trapezoidal method.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
μg*h/mL | 10.6 (2.67) | 11.3 (2.99)

6. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): Maximum Plasma Concentration (Cmax)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  Is defined Cmax the maximum observed concentration.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
μg/mL | 6.69 (1.88) | 7.97 (2.19)

7. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): Time to Maximum Plasma Concentration (Tmax)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  Is defined T max the time at which Cmax was apparent.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 12
h | 0.501 (0.00481) | 0.542 (0.144)

8. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): Half-life (t1/2)
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  Is defined T1/2 The apparent terminal half-life, calculated from Log e 2 / z.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 10
h | 3.77 (6.56) | 2.88 (1.40)

9. Primary Outcome: Change From Baseline in Area of Hyperalgesia (cm^2) Post-capsaicin Injection by MMRM Analysis. (Part B)
Description: The area of mechanical hyperalgesia was assessed using a standard 24 g von Frey hair. The von Frey hair was applied at 1-second intervals along each of the 4 lines intersecting at the injection site drawn onto the skin before the injection. Stimulation began distal from the injection site and advanced in 1 cm increments toward the injection site until a pain response was elicited. Subjects were asked to report when the von Frey hair first began to cause any pain sensation or discomfort and the distance of that point from the injection site in centimetres for each line at each timepoint was recorded.
Time Frame: Day 1 at 15, 30, 60, 90 and 120 minutes post injection
Population: Pharmacodynamic Set: PD Analysis Set consisted of all randomised subjects who received a dose of randomised therapy and were administered the ID capsaicin injection. This population was used for all PD analyses and PD analysis was performed by actual treatment received.
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
cm^2
  at 15 minutes post injection. The mean is an adjusted mean | 11.87 (6.37) | 4.95 (6.36) | 14.36 (6.38) | 8.76 (6.37) | 23.15 (6.37) | 5.41 (6.36) | 12.28 (6.37) | 11.85 (6.36)
  at 30 minutes post injection.The mean is an adjusted mean | 13.55 (6.81) | 4.12 (6.81) | 16.17 (6.84) | 14.73 (6.80) | 17.02 (6.82) | 5.69 (6.80) | 15.67 (6.81) | 1.45 (6.82)
  at 60 minutes post injection.The mean is an adjusted mean. | 12.16 (6.80) | 7.56 (6.80) | 16.31 (6.81) | 12.06 (6.80) | 12.89 (6.80) | -2.49 (6.80) | 6.28 (6.80) | 0.18 (6.81)
  at 90 minutes post injection.The mean is an adjusted mean. | 1.83 (6.34) | -6.64 (6.35) | 6.93 (6.35) | 7.38 (6.35) | 7.23 (6.34) | -4.23 (6.35) | 0.32 (6.35) | -0.51 (6.35)
  at 120 minutes post injection.The mean is an adjusted mean. | -0.42 (6.41) | -10.09 (6.44) | 9.64 (6.40) | 2.57 (6.41) | 2.40 (6.41) | -10.89 (6.42) | -8.22 (6.44) | -6.43 (6.40)
Statistical Analysis 1: Comparison: KLS 40 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.998, Mixed Model Repeated Measures; The p value was determined using MMRM model, based on treatment, timepoint, baseline value as covariable and subject as a random effect; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-17.81 to 17.86]
Statistical Analysis 2: Comparison: KLS 80 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.445, Mixed Model Repeated Measures. — The p value was determined using MMRM model, based on treatment, timepoint, baseline value as covariable and subject as a random effect; Mean Difference (Final Values) = -6.90, 95% CI 2-sided [-24.73 to 10.93]
Statistical Analysis 3: Comparison: KLS 160 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.781, Mixed Model Repeated Measures. — [p-value comment as in outcome 9, analysis 2]; Mean Difference (Final Values) = 2.51, 95% CI 2-sided [-15.33 to 20.36]
Statistical Analysis 4: Comparison: KLS 40 Mg-GABA 17 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.732, Mixed Model Repeated Measures. — [p-value comment as in outcome 9, analysis 2]; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-20.93 to 14.75]
Statistical Analysis 5: Comparison: KLS 80 mg- GABA 34 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.212, Mixed Model Repeated Measures. — [p-value comment as in outcome 9, analysis 2]; Mean Difference (Final Values) = 11.30, 95% CI 2-sided [-6.53 to 29.14]
Statistical Analysis 6: Comparison: KLS 160 Mg-GABA 68 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.476, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -6.44, 95% CI 2-sided [-24.27 to 11.39]
Statistical Analysis 7: Comparison: Gabapentin 300 mg (Part B) vs Placebo (Part B); Outcome Measure at 15 minutes post injection; Test type: Superiority; p = 0.962, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-17.40 to 18.26]
Statistical Analysis 8: Comparison: KLS 40 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.211, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 12.10, 95% CI 2-sided [-6.96 to 31.16]
Statistical Analysis 9: Comparison: KLS 80 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.782, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 2.67, 95% CI 2-sided [-16.40 to 21.73]
Statistical Analysis 10: Comparison: KLS 160 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.129, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 14.72, 95% CI 2-sided [-4.34 to 33.78]
Statistical Analysis 11: Comparison: KLS 40 Mg-GABA 17 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.171, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 13.27, 95% CI 2-sided [-5.80 to 32.35]
Statistical Analysis 12: Comparison: KLS 80 mg- GABA 34 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.108, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 15.56, 95% CI 2-sided [-3.49 to 34.62]
Statistical Analysis 13: Comparison: KLS 160 Mg-GABA 68 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.661, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 4.24, 95% CI 2-sided [-14.83 to 23.30]
Statistical Analysis 14: Comparison: Gabapentin 300 mg (Part B) vs Placebo (Part B); Outcome Measure at 30 minutes post injection; Test type: Superiority; p = 0.142, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 14.21, 95% CI 2-sided [-4.85 to 33.27]
Statistical Analysis 15: Comparison: KLS 40 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.216, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 11.98, 95% CI 2-sided [-7.08 to 31.04]
Statistical Analysis 16: Comparison: KLS 80 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.445, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 7.38, 95% CI 2-sided [-11.71 to 26.48]
Statistical Analysis 17: Comparison: KLS 160 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.096, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 16.13, 95% CI 2-sided [-2.92 to 35.19]
Statistical Analysis 18: Comparison: KLS 40 Mg-GABA 17 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.220, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 11.89, 95% CI 2-sided [-7.19 to 30.96]
Statistical Analysis 19: Comparison: KLS 80 mg- GABA 34 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.189, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 12.71, 95% CI 2-sided [-6.35 to 31.78]
Statistical Analysis 20: Comparison: KLS 160 Mg-GABA 68 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.782, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -2.67, 95% CI 2-sided [-21.75 to 16.41]
Statistical Analysis 21: Comparison: Gabapentin 300 mg (Part B) vs Placebo (Part B); Outcome Measure at 60 minutes post injection; Test type: Superiority; p = 0.528, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 6.10, 95% CI 2-sided [-12.98 to 25.18]
Statistical Analysis 22: Comparison: KLS 40 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.795, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [-15.45 to 20.12]
Statistical Analysis 23: Comparison: KLS 80 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.497, mean difference; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -6.13, 95% CI 2-sided [-23.96 to 11.69]
Statistical Analysis 24: Comparison: KLS 160 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.409, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 7.44, 95% CI 2-sided [-10.34 to 25.21]
Statistical Analysis 25: Comparison: KLS 40 Mg-GABA 17 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.382, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 7.89, 95% CI 2-sided [-9.92 to 25.70]
Statistical Analysis 26: Comparison: KLS 80 mg- GABA 34 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.390, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 7.74, 95% CI 2-sided [-10.05 to 25.54]
Statistical Analysis 27: Comparison: KLS 160 Mg-GABA 68 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.680, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -3.72, 95% CI 2-sided [-21.54 to 14.10]
Statistical Analysis 28: Comparison: Gabapentin 300 mg (Part B) vs Placebo (Part B); Outcome Measure at 90 minutes post injection; Test type: Superiority; p = 0.927, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-16.99 to 18.65]
Statistical Analysis 29: Comparison: KLS 40 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.508, Mixed Model Repeated Measures. — [p-value comment as in outcome 9, analysis 2]; Mean Difference (Final Values) = 6.02, 95% CI 2-sided [-11.95 to 23.98]
Statistical Analysis 30: Comparison: KLS 80 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.688, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -3.65, 95% CI 2-sided [-21.66 to 14.35]
Statistical Analysis 31: Comparison: KLS 160 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.079, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 16.08, 95% CI 2-sided [-1.88 to 34.03]
Statistical Analysis 32: Comparison: KLS 40 Mg-GABA 17 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.323, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 9.00, 95% CI 2-sided [-8.96 to 26.96]
Statistical Analysis 33: Comparison: KLS 80 mg- GABA 34 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.183, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 11.23, 95% CI 2-sided [-5.39 to 27.85]
Statistical Analysis 34: Comparison: KLS 160 Mg-GABA 68 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.756, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -2.61, 95% CI 2-sided [-19.24 to 14.02]
Statistical Analysis 35: Comparison: Gabapentin 300 mg (Part B) vs Placebo (Part B); Outcome Measure at 120 minutes post injection; Test type: Superiority; p = 0.638, Mixed Model Repeated Measures; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 3.96, 95% CI 2-sided [-12.68 to 20.59]

10. Primary Outcome: Plasma PK Concentrations and Parameters of Ketoprofen (Part A): AUC From Zero to Infinity (AUC0-∞),
Description: PK parameters of ketoprofen when administered alone and when administered in combination with gabapentin in healthy male subjects were assessed.
  AUC0-∞ - area under the concentration versus time curve from time zero to infinity The area under the concentration-time curve estimated from time zero to infinity as the sum of the two areas: AUC0-t and AUCextrap, where AUCextrap is calculated as Ct / z. Estimates will be considered to be unreliable if the extrapolated area (AUCextrap) is >20%.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | KLS 80 mg (Part A) | KLS 80 Mg-GABA 34 mg (Part A)
Number analyzed (Participants) | 12 | 10
μg*h/mL | 10.7 (2.96) | 11.4 (3.06)

11. Secondary Outcome: Adverse Events (Part A)
Description: An AE is any untoward medical occurrence in a study subject which either emerges or worsens from screening, during the clinical study, regardless of its potential relationship to the medicinal product. An AE, therefore, can be any unfavourable or unintended sign, including a clinically-significant abnormal laboratory finding, symptom, or disease temporally associated with the use of a medical product, whether or not it is considered to be study medication related.
  Data define number of AE reported; frequency for each AE not being reported. Please note: these data in the CSR, as per study crossover design, are provided "per sequence" and not "per intervention". Hence, their representation "per intervention" it's not applicable.
Time Frame: Through part A, from screening day up to 5 to 7 days post final dose, i.e. up to 7 weeks
Population: Safety Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS).
Measure: Number; unit: Number of events
Groups:
- "KLS 80 mg Alone, *Then* KLS 80 Mg and GABA 34 mg" (PART A): KLS 80 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules will be administered with 240 mL of water.
- "KLS 80 Mg and GABA 34 mg *Then* KLS 80 mg Alone" (PART A): KLS-GABA 80 mg-34 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules are administered with 240 mL of water.
  To maintain the blind, subjects assigned to receive 80 mg-34 mg KLS-GABA also receive a placebo capsule (dummy placebo).
Arm/Group | "KLS 80 mg Alone, *Then* KLS 80 Mg and GABA 34 mg" (PART A) | "KLS 80 Mg and GABA 34 mg *Then* KLS 80 mg Alone" (PART A)
Number analyzed (Participants) | 6 | 6
Number of events
  Overall TEAE | 2 | 1
  Serious treatment-emergent adverse event | 0 | 0
  TEAE Leading to Discontinuation | 0 | 0
  TEAE leading to Death | 0 | 0
  Treatment-emergent adverse event: Mild Severity | 2 | 1
  Treatment-emergent adverse event: Moderate Severity | 0 | 0
  Treatment-emergent adverse event: Severe Severity | 0 | 0
  TEAE: Not Related to Treatment | 2 | 0
  TEAE: Unlikely Related to Treatment | 0 | 1
  TEAE: Possibly Related to Treatment | 0 | 0
  TEAE: Probably Related to Treatment | 0 | 0
  TEAE: Definitely Related to Treatment | 0 | 0
  TEAE: Related to Treatment | 0 | 0

12. Secondary Outcome: Subjective Rating of Pain From the ID Capsaicin Model (Part B)
Description: Measurement of Pain Score (mm) Over Time. Pain is assessed through a visual analogue scale (VAS) consisting of a 100 mm line, with 0 representing "no pain'' and 100 "worst pain imaginable." Subjects are asked to mark the VAS using a single vertical stroke at the point they consider to appropriately reflect their level of pain from the injection of capsaicin (not general pain).
Time Frame: Prior to (within 15 minutes) and at the 15-, 30-, 60-, 90- and 120-minutes post-injection.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
score on a scale
  Pre-Capsaicin Injection | 0.44 (1.365) | 0.88 (2.125) | 0.69 (2.056) | 0.88 (2.918) | 0.06 (3.296) | 0.00 (3.055) | 0.44 (0.892) | 0.56 (3.425)
  15 Minutes Post Injection | -2.56 (15.849) | 3.25 (19.182) | -5.13 (12.638) | 3.63 (15.949) | -1.50 (14.320) | -3.75 (15.813) | -2.94 (13.542) | -6.81 (11.862)
  30 Minutes Post Injection | 21.94 (17.789) | 30.50 (21.891) | 29.38 (18.846) | 27.19 (17.848) | 23.13 (17.393) | 24.44 (15.349) | 29.44 (20.324) | 15.50 (13.866)
  60 Minutes Post Injection | 10.38 (9.351) | 15.06 (13.897) | 8.88 (7.338) | 10.88 (10.424) | 10.56 (13.171) | 8.88 (11.039) | 8.56 (9.598) | 5.25 (8.323)
  90 Minutes Post Injection | 2.75 (3.624) | 3.13 (4.801) | 2.56 (4.427) | 3.31 (3.911) | 3.69 (5.930) | 2.25 (3.066) | 2.81 (5.431) | 1.50 (2.683)
  120 Minutes Post Injection | 1.38 (2.446) | 1.75 (2.436) | 1.25 (1.807) | 1.88 (2.156) | 1.50 (2.422) | 1.00 (0.966) | 1.50 (4.163) | 0.44 (0.814)

13. Secondary Outcome: Change From Baseline of Pain Score of Hyperalgesia (NRS) by MMRM Analysis.(Part B)
Description: Pain reduction/analgesia is measured through visual analogue scale (VAS) consisting of a 100 mm line, with 0 representing "no pain'' and 100 "worst pain imaginable." Subjects are asked to mark the VAS using a single vertical stroke at the point they consider to appropriately reflect their level of pain from the injection of capsaicin (not general pain). A new VAS are provided for each time-point and subjects are not allowed to see their previous VAS responses. The VAS is scored by measuring from the left-hand end of the scale to the point where the subject has marked the line, and the distance in mm recorded.
Time Frame: Day 1 at 15, 30, 60, 90 and 120 minutes post injection
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
units on a scale
  15 Minutes Post Injection | 0.10 (0.37) | 0.94 (0.37) | 0.46 (0.37) | 0.81 (0.37) | 0.75 (0.37) | 0.79 (0.37) | 0.80 (0.37) | 0.01 (0.37)
  30 Minutes Post Injection | 0.05 (0.38) | 0.58 (0.39) | 0.30 (0.38) | 0.06 (0.39) | 0.47 (0.39) | 0.39 (0.38) | 0.46 (0.39) | -0.51 (0.38)
  60 Minutes Post Injection | -0.67 (0.32) | 0.00 (0.32) | -0.30 (0.32) | -0.50 (0.32) | 0.02 (0.32) | -0.18 (0.32) | -0.08 (0.32) | -0.49 (0.32)
  90 Minutes Post Injection | -0.68 (0.31) | -0.56 (0.31) | -0.25 (0.31) | -0.54 (0.31) | -0.24 (0.31) | -0.37 (0.31) | -0.23 (0.31) | -0.88 (0.31)
  120 Minutes Post Injection | -0.58 (0.30) | -0.79 (0.30) | -0.65 (0.30) | -0.59 (0.30) | -0.70 (0.30) | -0.33 (0.30) | -0.52 (0.30) | -0.92 (0.30)

14. Secondary Outcome: Change From Baseline of Area of Brush-evoked Allodynia From the ID Capsaicin Model (Part B)
Description: This outcome is assessed by sweeping a standard paintbrush at 1-second intervals across each of the 4 lines intersecting at the injection site drawn onto the skin before the injection. Stimulation begins distal from the injection site and advances in 1 cm increments toward the injection site until a pain response is elicited. Subjects are asked to indicate when the brush first begins to cause any pain or discomfort and the distance of that point from the injection site in centimetres for each line at each time-point is recorded. The area of allodynia was then calculated
Time Frame: Prior to (within 15 minutes) and at the 15-, 30-, 60-, 90- and 120-minutes post-injection.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
cm^2
  Pre-Capsaicin Injection | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  15 Minutes Post Injection | 4.574 (23.6690) | 1.769 (22.2854) | 4.087 (26.5438) | 11.246 (21.8903) | 0.375 (31.3485) | -4.861 (24.1747) | -4.083 (23.4260) | 2.011 (28.6385)
  30 Minutes Post Injection | 1.904 (29.8020) | -6.738 (20.1917) | 8.259 (22.2606) | 9.301 (28.4396) | 3.955 (28.6202) | -1.524 (26.5909) | -4.178 (23.6343) | -5.425 (34.2194)
  60 Minutes Post Injection | 4.176 (17.0876) | -5.060 (19.2494) | 5.878 (11.6536) | 8.264 (22.6764) | -2.630 (10.5206) | -6.056 (20.7553) | -11.710 (21.6124) | -4.641 (19.9627)
  90 Minutes Post Injection | 5.238 (12.8091) | -1.791 (9.5419) | 4.841 (10.5503) | 3.646 (17.8697) | -1.104 (12.9476) | -2.719 (16.2512) | 3.846 (16.6439) | -2.526 (11.6839)
  120 Minutes Post Injection | 0.641 (6.3370) | -4.752 (12.7411) | 3.206 (9.2605) | 5.978 (24.1098) | -0.813 (14.1667) | -0.596 (6.5890) | -0.023 (9.2870) | -5.349 (11.4016)

15. Secondary Outcome: Change From Baseline in Pain Score of Brush-evoked Allodynia From the ID Capsaicin Model (Part B)
Description: Change from Baseline of Pain in response to brush stimulation of the allodynic area is recorded using an 11-point NRS ranging from 0 ("no pain") to 10 ("worst possible pain"). The pain score reflects the maximum pain experienced during the assessment.
Time Frame: Prior to (within 15 minutes) and at the 15-, 30-, 60-, 90- and 120-minutes post-injection.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
score on a scale
  Pre-Capsaicin Injection | 0.06 (0.250) | 0.00 (0.365) | 0.00 (0.000) | 0.00 (0.000) | -0.13 (0.500) | -0.06 (0.250) | 0.00 (0.000) | 0.00 (0.000)
  15 Minutes Post Injection | -0.63 (0.806) | 0.19 (1.905) | -0.38 (1.147) | 0.19 (1.223) | -0.50 (1.033) | -0.25 (1.342) | -0.13 (0.885) | -0.56 (1.590)
  30 Minutes Post Injection | -0.19 (0.981) | -0.19 (1.276) | -0.50 (0.966) | 0.31 (0.946) | 0.00 (1.033) | -0.38 (1.784) | -0.06 (0.854) | -0.56 (1.413)
  60 Minutes Post Injection | -0.38 (0.885) | -0.19 (1.109) | -0.13 (0.719) | 0.25 (1.438) | 0.06 (1.289) | -0.44 (1.263) | -0.50 (1.366) | -0.19 (1.047)
  90 Minutes Post Injection | -0.31 (0.704) | 0.00 (0.730) | 0.13 (0.500) | 0.00 (1.095) | -0.31 (1.078) | -0.38 (1.258) | -0.63 (1.708) | -0.19 (1.047)
  120 Minutes Post Injection | -0.06 (0.443) | 0.13 (0.619) | 0.06 (0.574) | -0.25 (0.856) | -0.31 (1.138) | -0.06 (1.063) | -0.56 (1.263) | -0.31 (0.793)

16. Secondary Outcome: Change From Baseline in Area of Flare (AF) From the ID Capsaicin Model (Part B)
Description: The AF is determined by tracing the outline of visible skin reddening on to a sheet of acetate placed on the skin using a fine-tipped, permanent marker. The area is subsequently measured using planimetry and the results recorded in the CRF.
Time Frame: Day 1 Pre-Capsaicin Injection and at 15, 30, 60, 90 and 120 minutes post injection
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
cm2
  Pre-Capsaicin Injection | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  15 Minutes Post Injection | 3.77 (21.565) | 6.27 (11.905) | 9.19 (13.719) | 6.33 (17.756) | 10.09 (25.933) | 6.16 (12.363) | 6.86 (20.153) | 8.44 (16.814)
  30 Minutes Post Injection | 6.58 (20.856) | 7.36 (8.660) | 7.14 (12.503) | 5.24 (16.808) | 15.33 (14.637) | 10.82 (14.225) | 7.48 (14.857) | 6.63 (15.525)
  60 Minutes Post Injection | 6.07 (10.843) | 4.58 (12.976) | 5.12 (17.524) | 8.14 (8.159) | 8.89 (10.602) | 5.96 (11.399) | 7.88 (12.083) | 2.39 (14.813)
  90 Minutes Post Injection | 0.73 (1.360) | 3.34 (8.184) | -0.34 (2.138) | 0.78 (1.596) | 0.41 (2.573) | 0.02 (0.813) | -0.71 (3.328) | 1.48 (3.694)
  120 Minutes Post Injection | -0.06 (0.675) | 0.19 (0.512) | 0.14 (0.961) | 0.20 (1.191) | 0.17 (0.910) | 0.26 (0.530) | 0.09 (0.558) | 0.18 (0.872)

17. Secondary Outcome: Plasma PK Concentrations (Part B)
Description: Plasma concentration levels of ketoprofen and gabapentin in Part B of the study are summarised by timepoint.
Time Frame: At Day 1 predose, pre-capsaicin and 2 hours post capsaicin
Population: PK Analysis Set: consisted of all subjects who received a dose of the IMP (KLS-GABA or KLS) and had evaluable PK data. Data were below limit of quantification (Not Evaluable) for all the 000 data presented in the table.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16
ug/mL
  Gabapentin Concentration: Pre Dose | 000 (000) | 000 (000) | 000 (000) | 000 (000) | 000 (000) | 000 (000) | 000 (000)
  Gabapentin Concentration: Pre Capsaicin Injection | 000 (000) | 000 (000) | 000 (000) | 0.189 (0.0815) | 0.321 (0.1370) | 0.693 (0.2455) | 1.375 (0.5394)
  Gabapentin Concentration: 2h Post Injection | 000 (000) | 000 (000) | 000 (000) | 0.182 (0.0312) | 0.320 (0.0714) | 0.675 (0.1572) | 2.241 (0.7926)
  Ketoprofen Concentration: Pre Dose | 000 (000) | 000 (000) | 000 (000) | 000 (000) | 000 (000) | 000 (000) | 000 (000)
  Ketoprofen Concentration: Pre Capsaicin Injection | 2.224 (0.6594) | 5.278 (1.0825) | 10.748 (2.6576) | 2.526 (0.5912) | 5.024 (1.0030) | 11.259 (2.6875) | 000 (000)
  Ketoprofen Concentration: 2h Post Injection | 0.456 (0.1582) | 1.056 (0.3847) | 2.106 (0.6011) | 0.473 (0.1487) | 1.036 (0.4056) | 2.267 (0.7075) | 000 (000)

18. Secondary Outcome: Adverse Events (Part B)
Description: An AE is any untoward medical occurrence in a study subject which either emerges, or worsens from Screening, during the clinical study, regardless of its potential relationship to the medicinal product. An AE, therefore, can be any unfavourable or unintended sign, including a clinically-significant abnormal laboratory finding, symptom, or disease temporally associated with the use of a medical product, whether or not it is considered to be study medication related. Adverse events may include pre- or post-treatment events that occur as a result of Protocol- mandated procedures (i.e., invasive procedures, modification of subject's previous therapeutic regimen).
  Data define number of AE reported; frequency for each AE not being reported.
Time Frame: The specific period of time over which adverse events data were collected was from screening day up to 5 to 7 days post final dose, i.e. up to 6 weeks for Part B
Population: Safety Analysis Set consisted of all subjects who received a dose of the IMP (KLS, KLS-GABA, gabapentin, or placebo). Safety data were presented by actual treatment received.
Measure: Number; unit: Number of events
Arm/Group | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
Number of events
  treatment-emergent adverse event | 7 | 5 | 2 | 1 | 8 | 4 | 5 | 8
  Serious treatment-emergent adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE leading to discontinuation of treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Life-threatening Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE Leading to Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  treatment-emergent adverse event: Mild Severity | 7 | 5 | 2 | 1 | 7 | 4 | 5 | 7
  treatment-emergent adverse event: moderate Severity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  treatment-emergent adverse event: Severe Severity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  treatment-emergent adverse event: Not Related with treatment | 5 | 3 | 1 | 1 | 7 | 3 | 4 | 7
  treatment-emergent adverse event: Unlikely Related with treatment | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  treatment-emergent adverse event: Possibly Related with treatment | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  treatment-emergent adverse event: Probably Related with treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  treatment-emergent adverse event: Definitely Related with treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  treatment-emergent adverse event: Related with treatment | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse events data were collected was from screening day up to 5 to 7 days post final dose, *up to 7 weeks for Part A* and *up to 6 weeks for Part B*"
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. Data define number and frequency for each AE are reported. Please note: safety data in the CSR, as per study design, are provided per sequence (PART A) and not per intervention.
Groups:
- KLS 80 mg (PART A): KLS 80 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules will be administered with 240 mL of water.
  Ketoprofen Lysine Salt combined with Gabapentin: KLS-GABA (80 mg-34 mg) in Part A Ketoprofen Lysine Salt: KLS (80 mg) alone in each treatment period in Part A
- KLS 80 Mg and GABA 34 mg (PART A): KLS-GABA 80 mg-34 mg capsules are administered once in the morning of Day 1 in Part A in Treatment Periods 1 and 2 in the fasted state, according to the randomization schedule. Capsules are administered with 240 mL of water.
Arm/Group | KLS 80 mg (PART A) | KLS 80 Mg and GABA 34 mg (PART A) | KLS 40 mg (Part B) | KLS 80 mg (Part B) | KLS 160 mg (Part B) | KLS 40 Mg-GABA 17 mg (Part B) | KLS 80 mg- GABA 34 mg (Part B) | KLS 160 Mg-GABA 68 mg (Part B) | Gabapentin 300 mg (Part B) | Placebo (Part B)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12 | 6/16 | 3/16 | 2/16 | 1/16 | 6/16 | 4/16 | 5/16 | 6/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KLS 80 mg (PART A) (N=12) | KLS 80 Mg and GABA 34 mg (PART A) (N=12) | KLS 40 mg (Part B) (N=16) | KLS 80 mg (Part B) (N=16) | KLS 160 mg (Part B) (N=16) | KLS 40 Mg-GABA 17 mg (Part B) (N=16) | KLS 80 mg- GABA 34 mg (Part B) (N=16) | KLS 160 Mg-GABA 68 mg (Part B) (N=16) | Gabapentin 300 mg (Part B) (N=16) | Placebo (Part B) (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04802967/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT04802967/SAP_001.pdf